CLINICAL TRIAL: NCT02931396
Title: Functional Electrical Stimulation Use in Trans-tibial Amputations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alicia Koontz (Other)
Responsible Party: Sponsor-Investigator, Alicia Koontz, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO14050193
Record Dates: First submitted 2016-01-25; First posted 2016-10-13 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Traumatic Amputation of Lower Extremity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FES intervention (Experimental): Study participants who are randomized into the intervention group will be fitted with a portable commercially available surface FES device and instructed in its use by a study investigator. Participants will be directed to use the FES 30 minutes a day for the first week, one hour a day during the next week, 90 minutes a day during the third week, and then a minimum of 2 hours per day or 10 hours per week for the next three months at home.
  Interventions: Device: FES
- Control (No Intervention): Participants will be asked to continue their activities of daily living as usual.

INTERVENTIONS:
Device: FES
  Arms: FES intervention

SUMMARY:
The purpose of this study is to demonstrate the efficacy of functional electrical stimulation (FES) for trans-tibial amputees. The investigators aim to demonstrate that providing three months of FES intervention will increase knee extension strength, increase volume of the residual limb and decrease chronic and phantom pain.

DETAILED DESCRIPTION:
SUMMARY STUDY GOALS: The purpose of this study is to demonstrate the efficacy of FES for trans-tibial amputees. The investigators aim to demonstrate that providing three months of FES intervention will increase knee extension strength, increase volume of the residual limb and decrease chronic and phantom pain.

EXPERIMENTAL DESIGN: Randomized control trial METHODS: Twenty participants will be recruited and randomly divided into two groups, one group will receive the FES intervention while the other group will continue with activities of daily living. Both groups will keep a daily log of number of hours the prosthesis is worn, number of hours the FES is worn (if used) and any changes in skin conditions or medications. Both groups will return for assessment visits at 4, 8, and 12 weeks and a follow up visit 3 months post-intervention for investigators to inspect the residual limb and check the fit of the prosthetic socket, record residual limb knee extension strength on the Biodex machine, take measurements (circumferences and lengths) of the residual limb with a tape measure and ruler, scan the limb with the hand held three-dimensional motion-tracking laser scanner system and the participant will be asked to complete a pain questionnaire. The Prosthetic Evaluation Questionnaire (PEQ) will be completed at the 12 week and the 3 month follow-up visits. Although outcomes data were captured during each assessment visit (0, 4, 8 and 12 weeks and 3 months), changes in the primary outcomes (strength, volume and pain) at timepoints 0 weeks (pre-intervention) and 12 weeks (post- intervention) were of primary interest.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age.
* Participants have a unilateral trans-tibial amputation with a minimum of a 4" residual limb. This length of amputation was chosen to provide for adequate surface area for the electrodes.
* Participants must be a minimum of two years postoperative to insure proper healing of the limb has occurred.
* Participants have chronic limb pain.
* No prior experience in using TENS or FES.

Exclusion Criteria:

* No cardiac conditions, such as hypertension, congestive heart failure, or a pacemaker.
* People with severe diabetes who have insensate skin and or neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-02-03 (Actual); Study Completion 2018-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FES Intervention: Study participants who are randomized into the intervention group will be fitted with a portable commercially available surface FES device and instructed in its use by a study investigator. Participants will be directed to use the FES 30 minutes a day for the first week, one hour a day during the next week, 90 minutes a day during the third week, and then a minimum of 2 hours per day or 10 hours per week for the next three months at home.
  FES
Period: Overall Study
Arm/Group | FES Intervention | Control
Started | 10 | 10
Completed | 5 | 10
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FES Intervention | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (10.4) | 49.9 (16.8) | 52.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Extension Isometric Strength (Peak Torque) Using the Biodex Measurement System
Description: Residual limb knee extension isometric strength was tested using a standardized Biodex protocol and custom attachment. The lever arm of the Biodex was positioned at 60 degrees of knee flexion, with the support cushion modified for the amputee and positioned at the mid-tibia. The participant was asked to extend their knee against the arm as hard as they could for five seconds.
Time Frame: baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Nm/kg
Arm/Group | FES Intervention | Control
Number analyzed (Participants) | 5 | 10
Nm/kg | -0.1 [-6.0 to 5.7] | 2.2 [-1.4 to 5.8]
Statistical Analysis 1: Comparison: FES Intervention vs Control; Test type: Superiority; p = 0.768, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 2.3

2. Primary Outcome: Change in Residual Limb Volume Using 3-D Scanner
Description: 3-D motion-tracking laser scanning system was used to determine residual limb volume in cm
Time Frame: baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | FES Intervention | Control
Number analyzed (Participants) | 5 | 10
cm | -1.6 [-13.9 to 10.7] | 23.9 [-39.8 to 87.6]
Statistical Analysis 1: Comparison: FES Intervention vs Control; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 25.5

3. Primary Outcome: Change in Residual Limb Pain Using Likert Scale Pain Questionnaire
Description: Scores were reported on a 0 to 10 scale with higher scores representing higher pain levels
Time Frame: baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FES Intervention | Control
Number analyzed (Participants) | 5 | 10
units on a scale | -1.2 [-2.8 to 0.4] | 1.5 [-0.6 to 3.6]
Statistical Analysis 1: Comparison: FES Intervention vs Control; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 2.7

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | FES Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT02931396/Prot_SAP_000.pdf